CLINICAL TRIAL: NCT05184933
Title: Sleep and Circadian Mechanisms in Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Saurabh Thosar, Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00023776
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Cardiovascular Diseases; Cardiovascular Risk Factors; Circadian Rhythms; Sleep
Keywords: cardiovascular; circadian rhythms; sleep; blood pressure; constant routine; microneurography; hypertension; sleep regularization
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: All participants will complete all parts of the study. The order of completion of the second experiment (Overnight Sleep and Rested Wakefulness trials) will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dipping vs non-dipping HTN (Experimental): Participants will wear an ambulatory blood pressure monitor (SpaceLabs, Inc.) which will take their blood pressure in 20-30-minute intervals for 24-48 hours to determine blood pressure dipping status.
  All participants in this arm will complete the experiments in this order:
  1. At-home polysomnography;
  2. Constant Routine protocol;
  3. Rested Wakefulness Trial AND Overnight Sleep Trial (Randomized crossover);
  4. Sleep Regularization Trial
  Interventions: Other: At-home Polysomnography; Other: Circadian Protocol; Other: Rested Wakefulness Trial; Other: Overnight Sleep Trial; Behavioral: Regularized Sleep Schedule

INTERVENTIONS:
Other: At-home Polysomnography — Participants will complete one night of unattended polysomnography in their home environment (SOMNOtouch RESP, SOMNOmedics America Inc., FL, USA).
Other: Circadian Protocol — Participants will spend 4 days/3 nights in the laboratory to uncover circadian rhythms. After 2 nights for acclimatization and baseline measurements, participants will stay awake for 28 hours in dim light, constant temperature, and semi-recumbent posture. Participants will be provided with standardized snacks regularly. Polysomnography, core body temperature, sleep, finger oximetry, electrocardiogram (ECG), and beat-to-beat BP will (except microneurography) be measured throughout. Blood will be drawn every 2-4h to analyze catecholamines, renin activity, and aldosterone. All other measurements, including BP, heart rate (HR), and flow-mediated dilation will be performed regularly. Salivary samples will be collected every 2hrs (when awake) to analyze melatonin levels. A recovery sleep period will be provided and baseline testing procedures will be performed. Investigators may acquire direct recordings of sympathetic activity using microneurography.
  Other Names: Constant Routine
Other: Rested Wakefulness Trial — Participants will start wearing an ambulatory BP monitor upon admission. Participants will be instrumented with full polysomnography (except leg myogram), and an intravenous catheter will be placed in the non-dominant arm. Participants will receive a standardized snack, and dinner ~4 hours before the start of the trial. Participants will be instrumented for microneurography. Participants will be awake in bed in dim light (<8 lux). An investigator will constantly be present in the control room to monitor and ensure constant supine posture and wakefulness. Polysomnography, beat-by-beat BP, and neurogram for microneurography will be done throughout each trial into awakening; blood will be sampled before, during, and immediately after each trial (total of 8 samples in each trial). Flow-mediated dilation will be conducted before bed and after bed. The two trials will be conducted ~one month apart to accommodate the menstrual cycle phase in pre-menopausal females.
  Other Names: Randomized crossover with overnight sleep trial
Other: Overnight Sleep Trial — Participants will wear an ambulatory BP monitor upon admission. Participants will be instrumented with full polysomnography (except leg myogram), and an intravenous catheter will be placed in the non-dominant arm, and then participants will receive a standardized snack, and dinner 4 hours before the start of the trial. Polysomnography, beat-by-beat BP, and neurogram for microneurography will be done throughout each trial into awakening; blood will be sampled before, during, and immediately after each trial (total of 8 samples in each trial). Participants will be instrumented for microneurography. Participants will begin an 8-hour sleep opportunity (<0.1 lux) at their chosen sleep time. At the end of the sleep episode, participants will be gently awoken in a standardized fashion by use of a mild auditory stimulus. Flow-mediated dilation will be conducted before bed and after sleep. The two trials will be conducted one month apart to accommodate the menstrual cycle.
  Other Names: Randomized crossover with rested wakefulness trial
Behavioral: Regularized Sleep Schedule — All participants will be asked to maintain a self-selected bedtime (sleep duration not controlled) for two weeks as an intervention after the completion of the constant routine and both the resting wakefulness and overnight sleep trials. During this time, participants will be asked to call a time-stamped voicemail box upon waking and going to bed, as well as complete a daily sleep diary and wear an Actigraph device on their wrist. Ambulatory blood pressure will be measured at home before and at the end of the two-week intervention.

SUMMARY:
This study is a mechanistic clinical trial designed to investigate the effects of the circadian system and sleep on non-dipping blood pressure (BP) in people with hypertension (HTN).

DETAILED DESCRIPTION:
This study is a mechanistic clinical trial designed to study the effects of the circadian system and sleep on non-dipping blood pressure (BP) in people with hypertension (HTN). Investigators will study participants with dipping and non-dipping hypertension. All participants will partake in all experiments. First, investigators will assess sleep in the participants' home environment using unattended polysomnography. Participants will then complete a 5-day overnight forced desynchrony laboratory protocol to uncover circadian rhythms (Constant Routine). The second experiment is a randomized crossover protocol. Two trials (Overnight Sleep and Rested Wakefulness) will be completed in randomized order to separate the effects of sleep on non-dipping blood pressure while assessing nighttime cardiovascular mechanisms. Finally, investigators will pilot test if 2 weeks of sleep regularization impacts 24-hour BP.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-64
* BMI 18.5-42kg/m2
* Hypertension (average resting blood pressure between 130/80 mmHg and 160/100 mmHg)

Exclusion Criteria:

* Over 5 pack-years of smoking;
* Prior shift work within 12 months prior to the study;
* Travel greater than three time zones for at least 3 months;
* History of heart failure, cardiomyopathy, or history of bypass surgery, angioplasty, or previous myocardial infarction;
* Acute or chronic diseases (except hypertension) that may affect outcome measures;
* History of psychological conditions;
* Sleep disorders, like severe sleep apnea, insomnia, etc.;
* Prescription medications (Contraceptives and anti-hypertensive medications are permissible);
* History of Illicit drug use and alcohol dependency;
* 30 days free of cannabis use prior to the study;
* Pregnancy;
* Upper cut-off of 160/100 mmHg for BP

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Sleep duration (At-home Polysomnography) | 1-2 nights
  Sleep duration will be scored from the ActiGraph and correlated with the sleep and activity diary. Sleep duration measures the amount of time asleep (in minutes).
Sleep Episodes (At-home Polysomnography) | 1-2 nights
  Sleep episodes will be polysomnographically recorded and scored in 30-sec epochs for sleep stage, arousals, and respiratory events on SomnoMedics Domino Software. Values (based on software analysis) provide a description of what aspects of sleep are different between participants.
Blood pressure (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Blood pressure (BP; systolic and diastolic) will be measured in a supine or semi-recumbent position. Investigators will measure beat-by-beat BP using a noninvasive device employing the volume-clamp method with hydrostatic correction. Investigators will measure BP using a calibrated sphygmomanometer to record sporadic BP at regular intervals throughout the protocols. Investigators will study circadian rhythms in blood pressure between people with dipping vs non-dipping hypertension. Investigators will also study how overnight sleep affects blood pressure in these groups. Investigators will also study ancillary variables such as morning surge in blood pressure. All blood pressure measurements will be measured in mmHg.
Heart rate (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Heart rate will be measured in beats-per-minute (bpm). This is a standard marker of cardiovascular health.
Heart rate variability (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  For the duration of all in-laboratory studies, three channels of EKG are recorded (RA-V6) and stored at a sampling frequency of 256 Hz. This software will be used for peak detection (R-wave detection and subsequent heart rate variability (HRV) analysis to estimate cardiac vagal tone). Investigators will study circadian rhythms in heart rate between people with dipping vs non-dipping hypertension. Investigators will also study how overnight sleep affects heart rate variability in these groups. This is a measure of cardiac parasympathetic activity and cardiovascular health.
Epinephrine (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Plasma epinephrine (measured in plasma according to laboratory values) will be measured to estimate sympathetic output (stress). Higher values may indicate increased cardiovascular risk. Investigators will study circadian rhythms in Epinephrine between people with dipping vs non-dipping hypertension. Investigators will also study how overnight sleep affects Epinephrine in these groups.
Norepinephrine (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Plasma norepinephrine (measured in plasma according to laboratory values) will be measured to estimate sympathetic output (stress). Higher values may indicate increased cardiovascular risk. Investigators will study circadian rhythms in Norepinephrine between people with dipping vs non-dipping hypertension. Investigators will also study how overnight sleep affects Norepinephrine in these groups.
Aldosterone (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Plasma aldosterone (measured in plasma according to laboratory values) will be measured to estimate sympathetic output (stress). Higher values may indicate increased cardiovascular risk. Investigators will study circadian rhythms in Aldosterone between people with dipping vs non-dipping hypertension. Investigators will also study how overnight sleep affects Aldosterone in these groups.
Renin (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Plasma renin/activity (measured in plasma according to laboratory values) will be measured to estimate sympathetic output (stress). Higher values may indicate increased cardiovascular risk. Investigators will also study circadian rhythms in renin between people with dipping vs non-dipping hypertension. Investigators will also study how overnight sleep affects renin in these groups.
Vascular endothelial function (Circadian and Overnight sleep vs. rested wakefulness trial) | 7 days
  Investigators will measure endothelial function as flow-mediated dilation (FMD). Investigators will measure brachial artery FMD using standard procedures every 3 hours in the constant routine protocol and while awake during the overnight sleep vs. rested wakefulness trial. Investigators will also normalize FMD to the hyperemic shear. Investigators will study circadian rhythms in vascular function in people with dipping vs non-dipping hypertension. Investigators will also study if overnight sleep changes morning vascular function between these groups. Vascular function may be an indicator of cardiovascular health.
Magnitude of overnight blood pressure dipping (Overnight sleep vs. rested wakefulness trial) | 2 days
  Blood Pressure (BP) dipping will be calculated as the percent reduction in average nighttime BP reduction compared to daytime BP. Both systolic and diastolic blood pressure will be measured in mmHg. Blood pressure dipping status may be an indicator of cardiovascular health. Investigators will study whether being asleep or not changes the magnitude of dipping between dipping and non-dipping hypertension. Investigators will also measure ancillary variables such as average daytime BP, night time BP, and morning surge in BP.
Muscle sympathetic nerve activity (MSNA) (Overnight sleep vs. rested wakefulness trial and circadian trial) | 7 days
  MSNA may be directly measured by inserting a tungsten microelectrode (Frederick Haer, Bowdoinham, ME) into a peroneal nerve at the popliteal fossa. A reference electrode will be inserted subcutaneously 2-3 cm from the recording electrode. Both electrodes will be connected to a differential preamplifier and then to an amplifier to obtain mean voltage neurograms. Once investigators have confirmed a satisfactory post-ganglionic MSNA recording, the participants will be provided a 10 min non-recorded rest to ensure baseline levels. Data will be recorded using WinDaq/Pro data acquisition software (DATAQ Instruments, Akron, OH) and imported for analysis in the commercially available WinCPRS software program (Absolute Aliens; Turku, Finland). Investigators will also study how overnight sleep affects MSNA in these groups. Investigators may also study circadian rhythms in MSNA between people with dipping vs non-dipping hypertension.

SECONDARY OUTCOMES:
Ambulatory blood pressure (Sleep regularization trial) | 2 weeks
  Participants will be instructed to select a preferred bedtime time and ensure adherence to that time for 2-weeks. Investigators will not control sleep duration. After this trial, investigators will again measure 24-48 hour ambulatory BP. Both systolic and diastolic blood pressure will be measured in mmHg. Blood pressure dipping status will be assessed. BP dipping will be calculated as the percent reduction in average nighttime BP reduction compared to daytime BP. Blood pressure may be an indicator of cardiovascular health.
Blood pressure dipping status (Sleep regularization trial) | 2 weeks
  Participants will be instructed to select a preferred bedtime time and ensure adherence to that time for 2-weeks. Investigators will not control sleep duration. Both systolic and diastolic blood pressure will be measured in mmHg. Blood pressure dipping status will be assessed. BP dipping will be calculated as the percent reduction in average nighttime BP reduction compared to daytime BP. Blood pressure dipping status may be an indicator of cardiovascular health.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh S Thosar, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No